CLINICAL TRIAL: NCT04652258
Title: A Phase II, Open Label, Single Arm, Single Center Study to Evaluate Pyrexia Management (with or Without Any Other Cytokine Release Symptoms) Using Tocilizumab, an Humanized Monoclonal Antibody Against the Interleukin - 6 Receptor in BRAF+ Melanoma Patients Treated with Dabrafenib/ Trametinib +/- Immunotherapy
Brief Title: Pyrexia Management Using an IL-6 Antibody in BRAF+ Melanoma Patients Treated with Dabrafenib/ Trametinib +/- Immunotherapy
Acronym: Nov IIT- Pyrex
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: too few patients could be included
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NovartisIIT/ 2020-01929
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Pyrexia
MeSH Terms: conditions — Fever | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Other): The patients will be administered Tocilizmab (Actemra) at the following dosage :
  * First dose: 8mg/kg, max. 800mg iv. during 60min
  * If necessary second dose: 8mg/kg, max. 800mg iv. during 60min after 20-36 hours from first dose
  Interventions: Drug: Actemra

INTERVENTIONS:
Drug: Actemra — Dosage: 8mg/kg (max. 800mg) Actemra administered intravenously as an infusion over 60 min.

SUMMARY:
The study examines the development of fever after administration of Actemra (tocilizumab) in patients who have fever and other cytokine release symptoms (headache, nausea, palpitations, low blood pressure) due to cancer therapy (Tafinlar (dabrafenib) / Mekinist (trametinib) +/- immunotherapy) . The goal of the study is to better understand the side effects and to find an effective therapy against them.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent as documented by signature
2. Subjects (males and females) age ≥ 18 years
3. ECOG < 3
4. Subjects with pyrexia grade 1*- 4 and elevated CRP with persistent fever after one day of antipyretic therapy with or without at least one other additional symptom of cytokine release syndrome such as nausea, headache, tachycardia, hypotension, maculopapular rash, shortness of breath, transaminitis, renal failure, dehydration
5. Elevated CRP serum levels further than normal baseline levels (> 3.0 mg/L)
6. Subjects with resected, non-resectable, adjuvant or metastatic BRAF+ melanoma treated with :

   * BRAF inhibitor (dabrafenib) in combination with MEK inhibitor (trametinib)
   * BRAF inhibitor (dabrafenib) in combination with MEK inhibitor (trametinib) preceded by therapy with anti-PD-1/PD-L1 and/or anti CTLA-4 inhibitor
   * BRAF inhibitor (dabrafenib) in combination with MEK inhibitor (trametinib) plus anti-PD- 1/PD-L1 inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Pyrexia management | 1 hour to up to 72 hours.
  The primary outcome represents the proportion of patients that reduce to at least <38°C after tocilizumab infusion in BRAF+ melanoma patients under treatment with dabrafenib/trametinib +/- immunotherapy - pyrexia status will be assessed at screening visit and on every other defined visit until remission, by assessing body temperature.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Clinic of Dermatology, Zurich, Canton of Zurich, Switzerland